CLINICAL TRIAL: NCT07127341
Title: A Survey on the Use of Removable Functional Appliances Among Patients Undergoing Treatment at the Orthodontic Unit of Nice University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25Odonto05
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Orthodentic Appliances

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents of patient with removable functional appliance
  Interventions: Device: Patient with removable functional appliance

INTERVENTIONS:
Device: Patient with removable functional appliance — Survey (quiz) for patient who had malocclusion and/or a dysfunction treated removable functional appliance about the treatment, before, during and after treatment

SUMMARY:
The aim of the removable functional appliance is to restore functional balance (breathing, swallowing, chewing, etc.) and muscular balance (particularly of the facial muscles) in children. This contributes to the development of a harmonious and stable occlusion. This study aims to evaluate the level of cooperation, satisfaction, and perceived effectiveness of treatment among patients and their parents.The aim of this survey is to assess patient and parent cooperation, satisfaction, and perceived treatment effectiveness used for their neuromuscular, orthopedic, and dental effects of removable elastomeric appliances(orthodontic appliances, functional)."

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a malocclusion and/or a dysfunction which can be treated by removable functionnal appliance and their parents.

Exclusion Criteria:

* Patients who do not require functional education

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had a malocclusion and/or a dysfunction which can be treated by removable functionnal appliance and their parents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patient's satisfaction about the treatment removable functional appliance | A follow-up every 6 weeks for 6 months
  The satisfaction of patients is evaluated with a quiz (questionnaire) divided in three part : before, during and after treatment. ((34 questions quizz patient) with scale from 0 to 10 and free answers.
Evaluation of parent's satisfaction about the treatmtent with removable functional appliance | A follow-up every 6 weeks for 6 months
  The satisfaction of parents is evaluated with a quiz (questionnaire) divided in three part : before, during and after treatment. 25 questions quizz parents with scale from 0 to 10 and free answers.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France